CLINICAL TRIAL: NCT04058808
Title: Motivational Support for Patients With Atrial Fibrillation to Promote Weight Loss
Brief Title: MOTIVATE AF Motivational Support for Patients With Atrial Fibrillation to Promote Weight Loss
Acronym: MOTIVATE AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CD19/124451
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with Atrial Fibrillation attending the clinic. (Experimental)
  Interventions: Other: Weight Watchers; Other: Slimming world; Other: Leeds 'One You'; Other: NHS Choices; Other: 5:2 diet; Other: Individuals own personal plan

INTERVENTIONS:
Other: Weight Watchers — online or in a weekly wellbeing workshop, there is a fee of £12.95 per month, this is a healthy lifestyle programme based on food items having a point attached to them depending on the calorie, fat and sugar content. Each member has a specific number of points per day to use on their meals. The healthier foods have fewer points therefore you can eat more of them.
Other: Slimming world — online or in a weekly class, there is a fee of £5 per week. Free foods can be consumed freely are low fat healthy options, healthy extras (bread/milk/pulses) can be consumed in moderation. Higher fat, higher calorific foods have a number of SYNS attached, each person has a set number of SYNS (sins) per week to use as they wish.
Other: Leeds 'One You' — a free weekly 1 hour class (run in various places across Leeds), a variety of topics are covered, from food labels to the Eat well guide. This eating plan is based on calorie counting.
Other: NHS Choices — a free on line programme that is based on restricting calories using the Eat well guide and encouraging physical activity.
Other: 5:2 diet — 5 days of eating normal calories (2000 Female, 2500 Male) and 2 days eating restricted 500 calories (this may be amended depending on the patient).
Other: Individuals own personal plan — the participant will explain in detail their own designed plan and this will be documented on the paper records.

SUMMARY:
This study is designed to look at the impact that support and motivation has on patients with Atrial Fibrillation's ability to lose weight and maintain this. We believe that weight loss has a positive impact on the reduction of symptoms of atrial fibrillation and can decrease the likelihood of the arrhythmia returning following cardio version.

This study is designed for patients who have a diagnosis of Atrial Fibrillation and have a Body Mass Index greater than 27.

In the study, we plan to provide support and motivation to patients with atrial fibrillation to encourage weight loss. There are several weight loss strategies available to follow. Information will be provided about each strategy to encourage informed choices. If the initial strategy chosen is not working, this can be change to a more suitable one as required. Follow up will be by telephone at 2 and 4 weeks then every month thereafter where you will be asked your weight and to clarify the weight loss strategy you are following. You will be seen at 6 and 12 months where you will have an ECG, BP check and your weight measured. A final telephone assessment will take place at 24 months.

We hope that the research will in the future help patients with Atrial Fibrillation manage and maintain their weight loss to improve their symptoms and prevent recurrence of the arrhythmia. The results of this study could potentially change practice in our centre by providing more structured weight loss clinics for patients with Atrial Fibrillation

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* BMI>27
* Symptomatic AF
* Committed to monthly follow up phone calls and bi annual visits.

Exclusion Criteria:

* Any co morbidity that would reduce life expectancy to within the year.
* Unable to commit to follow up.
* Patients recruited to weight loss studies that are on going

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Weight loss of at least 3% at end of year 1 | 1 year
  Participant has lost weight at end of year 1. (The weight loss is graded <3%, 3-10%, .10%)

IPD SHARING:
Plan to Share IPD: No